CLINICAL TRIAL: NCT03571373
Title: Paediatric Inflammatory Bowel Diseases Network for Safety, Efficacy, Treatment and Quality Improvement of Care: The PIBD-NET Inception Cohort and Safety Registry
Brief Title: PIBD-SETQuality: the Inception Cohort and Safety Registry
Acronym: PIBD-SETQ
Status: Recruiting | Type: Observational
Sponsor: PIBD-Net (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: PIBD-Net 2016-02
Record Dates: First submitted 2018-06-14; First posted 2018-06-27 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Only in a subgroup of all patients (n=300), in specific centers, serum, stool and biopsies of (un)affected tissue of the ileum and/or colon will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention due to the observational set-up of this study.

SUMMARY:
The purpose of this study is to analyse effectiveness and safety signals of current treatment strategies in routine practice for patients with pediatric-onset inflammatory bowel disease (PIBD) and to correlate this to their individual risk factors.

DETAILED DESCRIPTION:
In this prospective observational study children with newly diagnosed inflammatory bowel disease (IBD) will be included in the inception cohort. The primary aim of the inception cohort is to analyse the effectiveness and safety signals of current treatment strategies and to correlate them to individual risk factors. In order to capture information on rare and severe complications in PIBD as well, the safety registry was designed to estimate incidence and prevalence rates of these complications and get more insight in disease and treatment characteristics of these patients.

ELIGIBILITY:
Inclusion Criteria Inception cohort:

Newly diagnosed patient, <18 years of age, with a likely diagnosis of IBD or a confirmed diagnosis of IBD can be included in the study. In order to be eligible to continue in the study the subject must meet all of the following criteria:

* Diagnosis is based on history, physical examination, laboratory, endoscopic, radiological and histological features according to the revised Porto criteria (1)
* Diagnosis has been made or is confirmed within 2 months of inclusion
* Data on all diagnostic procedures are available for inclusion in the database
* Informed consent of patient (if indicated) and parents has been obtained
* Concerning the patients of whom biological specimens will be included: patients have not started IBD treatment yet

Inclusion Criteria Safety Registry:

Any child with IBD <19 years old with complications as detailed in the agreed safety monitoring list (or future updates of the list of conditions) can be reported. For the initial reporting of incident cases no patient identifiable details will be required.

Exclusion Criteria Inception cohort:

* Inability to read and understand the patient and family information sheets (for example insufficient knowledge of national language, where no health advocate or family member is available to translate and ensure full understanding of the study)
* Informed consent of patient or parents has not been obtained when required
* Patients on similar treatments as for IBD but for other conditions, or known with conditions directly affecting the IBD (e.g. immunodeficiency or major gastrointestinal resections)

Exclusion Criteria Safety registry: none.

Ages: 0 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with paediatric-onset IBD (either Crohn's disease, ulcerative colitis or IBD-unclassified).
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictors for outcome and treatment response or non-response | Over a period of three years after inclusion of the last patient.
  Factors predictive for outcome and treatment response or non-response This includes factors at baseline and 12 weeks after disease-onset that predict adverse outcomes (e.g. fibrostricturing disease, penetrating disease, active perianal fistula or abcess and need of surgery).

SECONDARY OUTCOMES:
New biomarkers as classifiers of response or non-response to therapy | Over a period of three years after inclusion of the last patient.
  Part of the children in the inception cohort will deliver biological specimens to develop new biomarkers as classifiers of disease risk of complicated disease or side effects in PIBD patients, as well as predictors of (non-)response to a specific immunomodulator or biological agent.
Identification of patients with rare and serious complications | Until the end of patients recruitment, for a period of 2 years.
  Secondary outcome is to identify patients with rare and serious complications of PIBD or its treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lissy de Ridder, MD, PhD, Principal Investigator — Erasmus MC-Sophia Children's Hospital; Nicholas Croft, MD, PhD, Principal Investigator — Barts and the London School of Medicine, Queen Mary University of London
Locations (2):
- Erasmus MC - Sophia Children's Hospital, Rotterdam, Netherlands
- Royal Hospital London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Timmer A, Behrens R, Buderus S, Findeisen A, Hauer A, Keller KM, Kliemann G, Lang T, Lohr W, Rzehak P, Koletzko S; CEDATA-GPGE Study Group. Childhood onset inflammatory bowel disease: predictors of delayed diagnosis from the CEDATA German-language pediatric inflammatory bowel disease registry. J Pediatr. 2011 Mar;158(3):467-473.e2. doi: 10.1016/j.jpeds.2010.09.014. Epub 2010 Nov 4. PMID 21051046
- [Background] De Greef E, Hoffman I, Smets F, Van Biervliet S, Bontems P, Hauser B, Paquot I, Alliet P, Arts W, Dewit O, De Vos M, Baert F, Bossuyt P, Rahier JF, Franchimont D, Vermeire S, Fontaine F, Louis E, Coche JC, Veereman G; IBD working group of BESPGHAN, BIRD. Paediatric Crohn Disease: Disease Activity and Growth in the BELCRO Cohort After 3 Years Follow-up. J Pediatr Gastroenterol Nutr. 2016 Aug;63(2):253-8. doi: 10.1097/MPG.0000000000001132. PMID 26835906
- [Derived] Nugteren S, Simons-Oosterhuis Y, Menckeberg CL, Hulleman-van Haaften DH, Lindenbergh-Kortleve DJ, Samsom JN. Endogenous secretory leukocyte protease inhibitor inhibits microbial-induced monocyte activation. Eur J Immunol. 2023 Feb;53(2):e2249964. doi: 10.1002/eji.202249964. Epub 2022 Dec 22. PMID 36480463
- [Derived] Aardoom MA, Kemos P, Tindemans I, Aloi M, Koletzko S, Levine A, Turner D, Veereman G, Neyt M, Russell RK, Walters TD, Ruemmele FM, Samsom JN, Croft NM, de Ridder L; PIBD-SETQuality consortium and PIBD-NET. International prospective observational study investigating the disease course and heterogeneity of paediatric-onset inflammatory bowel disease: the protocol of the PIBD-SETQuality inception cohort study. BMJ Open. 2020 Jul 1;10(7):e035538. doi: 10.1136/bmjopen-2019-035538. PMID 32611739